CLINICAL TRIAL: NCT03987945
Title: Prognostic Implications of Left Atrial Appendage Occlusion in Patients With Non-valvular Atrial Fibrillation at Shanghai Tenth People's Hospital
Brief Title: Left Atrial Appendage Occlusion in Patients With Non-valvular Atrial Fibrillation From Shanghai
Acronym: LAAO-SH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Other Study IDs: LAAO-SH
Record Dates: First submitted 2019-06-14; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Occlusion
Keywords: atrial fibrillation; left atrial appendage occlusion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Left atrial appendage occlusion: Patients with non-valvular atrial fibrillation who have received left atrial appendage occlusion procedure.
  Interventions: Device: left atrial appendage occlusion devices

INTERVENTIONS:
Device: left atrial appendage occlusion devices — All NVAF patients who are admitted for receiving left atrial appendage occlusion procedure, including Watchman, LAmbre, Lefort, and Leftear deveices.

SUMMARY:
The prognostic implication of left atrial appendage occlusion (LAAO) procedure in non-valvular atrial fibrillation (NVAF) patients from China is still unclear. We aim to investigate the impact of LAAO procedure on subsequent clinical outcomes in patients from China.

DETAILED DESCRIPTION:
Although the left atrial appendage occlusion (LAAO) procedure has increasingly been performed to prevent the occurrence of ischemic stroke events among patients with non-valvular atrial fibrillation (NVAF), the clinical benefits and prognostic implications of which have not been well characterized in patients from China. As a result, we aim to conduct an observational study to explore the prognostic impact of LAAO in patient with NVAF who are hospitalized in Shanghai Tenth People's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were admitted for NVAF undergoing LAAO procedure between January 2014 and December 2017 in the Cardiology Department of Shanghai Tenth People's Hospital;
* Adult patients (>18 years old).

Exclusion Criteria:

* Patients with rheumatic valvular disease;
* Patients with sick sinus syndrome;
* Patients who had a history of cardiac surgery (i.e., CABG);
* patients who had received the catheter radiofrequency ablation procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with NVAF who are referred for LAAO procedure.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebral events (MACCE) | From the time of performing LAAO procedure until occurrence of an outcome of interest, death, lose to follow up or Jan, 2020, maximum up to 6 years
  A composite of all-cause death, ischemic stroke, heart failure rehospitalization and major bleeding events

SECONDARY OUTCOMES:
All-cause death | From the time of performing LAAO procedure until occurrence of death, lose to follow up or Jan, 2020, maximum up to 6 years
  Death from any cause
Cardiovascular death | From the time of performing LAAO procedure until occurrence of death, lose to follow up or Jan, 2020, maximum up to 6 years
  Death from cardiovascular causes
Ischemic stroke | From the time of performing LAAO procedure until occurrence of an outcome of interest, death, lose to follow up or Jan, 2020, maximum up to 6 years
  Ischemic stroke is defined as the presence of a new focal neurologic deficit thought to be ischemia in origin, with signs or symptoms lasting>24h
Major bleeding | From the time of performing LAAO procedure until occurrence of an outcome of interest, death, lose to follow up or Jan, 2020, maximum up to 6 years
  The incidence of major bleeding as defined by BARC (3-5)
Heart failure rehospitalization | From the time of performing LAAO procedure until occurrence of an outcome of interest, death, lose to follow up or Jan, 2020, maximum up to 6 years
  Rehospitalization for heart failure
Pericardial effusion | From the time of performing LAAO procedure until occurrence of an outcome of interest, death, lose to follow up or Jan, 2020, maximum up to 6 years
  Pericardial effusion validated by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, M.D., Ph.D., Principal Investigator — Department of Cardiology, Shanghai Tenth People's Hospital
Locations (1):
- Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided